CLINICAL TRIAL: NCT03709108
Title: Safety and Feasibility of an Insulin Sensitivity-Informed Bolus Calculator in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Chiara Fabris, PhD, Research Associate, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 21040
Record Dates: First submitted 2018-10-08; First posted 2018-10-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Continuous Glucose Monitor; Insulin Sensitivity; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental-Control (Other): Subjects randomized to this Arm would go through the Experimental Admission (SI-informed bolus calculator) first and Control Admission (regular bolus calculator) second
  Interventions: Other: SI-Informed Bolus Calculator
- Control-Experimental (Other): Subjects randomized to this Arm would go through the Control Admission (regular bolus calculator) first and Experimental Admission (SI-informed bolus calculator) second
  Interventions: Other: SI-Informed Bolus Calculator

INTERVENTIONS:
Other: SI-Informed Bolus Calculator — The SI-Informed Bolus Calculator will be used to dose the dinner meal insulin bolus during the Experimental Admission

SUMMARY:
This is a single-center randomized crossover trial. The investigators will target completion of 15 adults (age 18-65 years) with Type 1 Diabetes who use an insulin pump. After completion of the Screening Visit, each subject will participate in a 28-day at home Data Collection Period while using their personal insulin pump, a personal glucometer, a study CGM, and a study activity tracker (i.e., Fitbit). This data collection period may be extended to obtain to gather more days of quality data, if needed per principal investigator judgement.

Once the data has been collected and processed, subjects will participate in two 24-hour admissions (Experimental and Control Admission) in a semi-controlled environment (i.e., hotel), performed in the assigned random order. During both admissions, subjects will use the personal insulin pump and glucometer, and a study CGM. The exercise session will consist of three 15-minute bouts of moderate-intensity exercise (i.e., stationary bicycle). Subjects will be provided a controlled dinner; the SI-informed bolus calculator will be used in the Experimental Admission while standard therapy will be used in the Control Admission. Subjects will then be observed overnight and discharged in the following morning.

DETAILED DESCRIPTION:
Individuals with Type 1 Diabetes (T1D) require exogenous insulin to keep their blood glucose concentration in a safe euglycemic range, because of the absent internal insulin secretion caused by the autoimmune destruction of pancreatic beta-cells. As a consequence, the quality of glycemic control in T1D is heavily dependent on multiple daily treatment decisions by the patients, which are complicated by a wide variety of factors influencing insulin demand (e.g., circadian rhythms, physical activity, food, stress, etc.). Insulin sensitivity (SI) is a key metabolic parameter in diabetes as it informs on how sensitive the body is to the effects of insulin. In general, if someone has higher SI, the amount of insulin required to lower his blood glucose levels is smaller than that needed by someone who has low sensitivity. However, SI levels within the same person are not constant, and fluctuations of SI happen very frequently in the life of subjects with diabetes, making insulin dosing very difficult to tune.

In this context, the aim of this research project is to develop an SI-informed insulin bolus calculator, with the aim of tailoring the insulin dose to the individual's insulin need at the time the bolus is administered. The SI-informed bolus calculator relies on a Kalman filter-based algorithm which uses continuous glucose monitoring (CGM) data, insulin, and meal records to estimate SI. For each subject, a 24-hour SI profile is computed using data collected over several days of monitoring, and the optimal bolus is then computed by adjusting the standard insulin dose by the ratio between usual SI (from the profile) and real-time SI of the individual at the time the bolus is administered. In this way, if the real-time SI is larger/smaller than the profile SI at that time of day, the insulin dose will be reduced/incremented accordingly.

The study is thus designed as a single-center randomized clinical trial targeting completion of 15 subjects, who will undergo a 28-day at home Data Collection Period followed by two 24-hour admissions (Control and Experimental Admission) performed in random order in a semi-controlled environment (i.e., hotel). The Data Collection is meant to collect data needed to build the 24-hour SI profile for the subject. During the admissions, subjects will undergo a 45-minute afternoon exercise session designed to alter the late-afternoon/evening SI. The dinner meal will then be controlled, and the postprandial glycemic control obtained using the standard bolus calculator (Control Admission) will be compared to the control obtained in response to the optimized SI-informed bolus calculator (Experimental Admission). Metrics computed on CGM data will be compared between the two admissions, including mean blood glucose, time above 250 and 300 mg/dL, time below 70 and 54 mg/dL, and time in 70-180 mg/dL, the primary outcome being the postprandial exposure to hypoglycemia as measured by the Low Blood Glucose Index (a glycemic variability indicator which summarizes the number and extent of low blood glucose events in one single number). If successful, this study will provide a novel, data-oriented paradigm for insulin dosing in T1D.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes for at least 12 months
2. Current use of an insulin pump for at least 12 months
3. Current or historical use of a CGM system for at least 6 months
4. Age ≥18 to ≤65 years old
5. HbA1c <8.5% at screening; if HbA1c <6.0% then total daily insulin must be ≥0.5 U/kg
6. For females, not currently known to be pregnant. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative urine pregnancy test will be required for all premenopausal women who are not surgically sterile. Subjects who become pregnant will be discontinued from the study
7. Willingness to use the same set of insulin therapy parameters (i.e., basal rate, insulin-to-carbohydrate ratio, correction factor) during both admissions
8. Willingness to upload data during the study
9. An understanding of and willingness to follow the protocol and sign the informed consent

Exclusion Criteria:

1. Diabetes ketoacidosis (DKA) in the 6 months prior to enrollment
2. Clinically significant electrocardiogram (ECG) found at Screening as determined by the study medical physician
3. Severe hypoglycemia resulting in seizure or loss of consciousness in the 6 months prior to enrollment
4. Currently being treated for a seizure disorder
5. Coronary artery disease or heart failure, unless written clearance is received from a cardiologist or primary care provider and documentation of a negative stress test within the year
6. History of cardiac arrhythmia (except for benign premature atrial contractions and benign premature ventricular contractions which are permitted)
7. Cystic fibrosis
8. Pregnancy, breast-feeding, or intention of becoming pregnant over time of study procedures
9. Abnormal liver function test results (Transaminase >2 times the upper limit of normal)
10. Abnormal renal function test results (calculated GFR <60 mL/min/1.73m2)
11. Uncontrolled thyroid disease (TSH undetectable or >10 mIU/L)
12. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:

    * Inpatient psychiatric treatment in the past 6 months for either the subject or the subject's care companion
    * Presence of a known adrenal disorder
    * Active gastroparesis
    * If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
13. Abuse of alcohol or recreational drugs
14. Infectious process not anticipated to resolve prior to study procedures (e.g. meningitis, pneumonia, osteomyelitis)
15. Uncontrolled arterial hypertension (Resting diastolic blood pressure >90 mmHg and/or systolic blood pressure >160 mmHg)
16. A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the protocol
17. Basal Rate <0.01 units/hour
18. Inability to be physically active for more than 30 minutes per day
19. Conditions that would make use of a CGM difficult (e.g., blindness, severe arthritis, immobility)
20. Current enrollment in another intervention clinical trial

List any restrictions on use of other drugs or treatments:

1. Medications being taken to lower blood glucose, such as Pramlintide, Metformin, GLP-1 Analogs such as Liraglutide, and nutraceuticals intended to lower blood glucose
2. Any other medication that the investigator believes is a contraindication to the subject's participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility of the SI-informed bolus calculator: Low Blood Glucose Index | LBGI will be assessed in the postprandial period following the controlled dinner meal (up to 4 hours following dinner) and overnight (e.g., from 11PM until 6AM), and will be compared between the two admissions.
  Safety and feasibility of the SI-informed bolus calculator as measured by overall and postprandial occurrence of hypoglycemia quantified using the Low Blood Glucose Index (LBGI) computed from CGM data. LBGI is a previously introduced glucose variability measure and strong predictor of severe hypoglycemia, designed to aggregate the frequency and extent of low blood glucose events into a single number. By this definition, a higher LBGI may indicate a large number of mild hypoglycemic events, a small number of significant events, or a combination of both. As a higher LBGI indicates higher exposure to hypoglycemia, LBGI is expected to be better (i.e., lower) when the optimized bolus calculator is used, as compared to standard therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Fabris, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fabris C, Nass RM, Pinnata J, Carr KA, Koravi CLK, Barnett CL, Oliveri MC, Anderson SM, Chernavvsky DR, Breton MD. The Use of a Smart Bolus Calculator Informed by Real-time Insulin Sensitivity Assessments Reduces Postprandial Hypoglycemia Following an Aerobic Exercise Session in Individuals With Type 1 Diabetes. Diabetes Care. 2020 Apr;43(4):799-805. doi: 10.2337/dc19-1675. Epub 2020 Mar 6. PMID 32144167

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT03709108/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT03709108/ICF_001.pdf